CLINICAL TRIAL: NCT00940160
Title: A Randomized, Double Blind, Placebo Controlled, Study To Compare The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Multiple Doses Of Intravenous Administration Of QAX576 In Controlled Or Partially Controlled Asthma Patients
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of QAX576 in Asthma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQAX576A2107
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2010-01

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- QAX576 1 mg/kg (Active Comparator)
  Interventions: Drug: QAX576
- QAX576 3 mg/kg (Active Comparator)
  Interventions: Drug: QAX576
- QAX576 10 mg/kg (Active Comparator)
  Interventions: Drug: QAX576
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAX576
  Arms: QAX576 1 mg/kg
Drug: QAX576
  Arms: QAX576 3 mg/kg
Drug: QAX576
  Arms: QAX576 10 mg/kg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is designed to investigate the safety and tolerability of multiple doses of QAX576 in controlled or partially controlled asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking male and female subjects age 18 to 65 years, inclusive; with controlled or partially controlled asthma who are otherwise healthy as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening. Female subjects are allowed to participate in this study if they are postmenopausal or surgically sterilized.
* Controlled or partially controlled asthma as defined in GINA 2007.
* At Screening, and Baseline, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed after the subject has rested for at least three (3) minutes.
* Female subjects must be post-menopausal as confirmed by FSH ≥ 40, or have been surgically sterilized at least 6 months prior to screening.
* Subjects must have a body mass index (BMI) within the range of 18 to 30 kg/m2.
* Male subjects must be using two methods of contraception, i.e., spermicidal gel plus condom, for the entire duration of the study, up to Study Completion visit, and refrain from fathering a child in the six (6) months after study completion

Exclusion criteria

* Smokers (use of tobacco products in the previous 3 months).
* Use of any prescription drugs other than stable (4 weeks) use of hormone replacement or thyroid replacement within four (4) weeks prior to dosing (other than medication required for treatment of asthma).
* Use of any over the counter (OTC) medication within forty eight (48) hours prior to dosing.
* Use of oral steroids within 12 weeks prior to dosing.
* Patients who have received an investigational drug in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulations, and for any other limitation of participation based on local regulations.
* Any immunotherapy with systemic biologics as a treatment therapy or during a clinical study with in the last 6 months.
* Any immunotherapy with subcutaneous injections for allergy (allergy shots), within 3 months.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to first dosing, or longer if required by local regulation.
* Patients suffering from hay fever at screening or likely to require treatment during the study.
* History of chronic respiratory disease other than asthma or chronic allergic rhinitis.
* Hospitalization for asthma in the last year.
* History of intubation/assisted ventilation for asthma in the last 5 years.
* History of autonomic dysfunction (e.g. history of fainting, orthostatic hypotension).
* History or presence of any surgical or medical condition or clinically significant abnormal laboratory findings, which, in the opinion of the investigator, may jeopardize the subject in case of participation in the study.
* History of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations.
* History of clinical schistosomiasis or travel within the preceding 6 months to an area with endemic schistosomiasis, including but not limited to Southeast Asia and Northwest Africa.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Measure: Assessing and comparing the safety and tolerability of multiple doses of QAX576 in controlled and partially controlled asthma patients. | 120 Days

SECONDARY OUTCOMES:
Assessing the pharmacokinetics of multiple doses of QAX576 in asthmatics | 120 Days
Assessing the effect of QAX576 on asthma control using assessments such as exhaled NO, FEV1 variability data captures by PIKO-1 home monitoring device and the extent of inhaled salbutamol use as rescue medication. | 120 Days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Russia (2):
  - Novartis Investigator Site, Moscow
  - Novartis Investigator Site, Saint Petersburg
- Novartis Investigator Site, Manchester, United Kingdom

REFERENCES:
- See also: Results for CQAX576A2107 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5704